CLINICAL TRIAL: NCT03195478
Title: A Phase 1/2 Study of Nivolumab (BMS-936558) in Combination With Ipilimumab (BMS-734016) in Chinese Participants With Previously Treated Metastatic or Recurrent Solid Tumors
Brief Title: A Study of Nivolumab in Combination With Ipilimumab in Chinese Participants With Previously Treated Advanced or Recurrent Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CA209-672
Record Dates: First submitted 2017-06-20; First posted 2017-06-22 (Actual); Results first posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-08

CONDITIONS: Solid Tumor
MeSH Terms: interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Nivo/Ipi Combination Therapy A (Experimental)
  Interventions: Drug: Nivolumab; Drug: Ipilimumab
- Nivo/Ipi Combination Therapy B (Experimental)
  Interventions: Drug: Nivolumab; Drug: Ipilimumab
- Nivo/Ipi Combination Therapy C (Experimental)
  Interventions: Drug: Nivolumab; Drug: Ipilimumab
- Nivo/Ipi Combination Arm D (Experimental)
  Interventions: Drug: Nivolumab; Drug: Ipilimumab

INTERVENTIONS:
Drug: Nivolumab — Specified dose on specified days
  Other Names: BMS-936558; Opdivo
Drug: Ipilimumab — Specified dose on specified days
  Other Names: BMS-734016; Yervoy

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of Nivolumab in combination with Ipilimumab in Chinese participants with previously treated late stage cancer.

ELIGIBILITY:
Inclusion Criteria:

* Mainland Chinese participants with advanced or recurrent solid tumors
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* One prior anti-cancer therapy that did not work or documented refusal to receive chemotherapy or biological therapy

Exclusion Criteria:

* Cancer that has spread to the brain or central nervous system unless it has been adequately treated . In addition, either no longer receiving corticosteroids, or on a stable or decreasing dose of no more than 10 mg daily prednisone (or equivalent)
* Active, known or suspected autoimmune disease or infection
* Positive blood screen for chronic infection of hepatitis B or hepatitis C (HCV antibody positive unless HCV RNA is negative)
* Prior immuno-oncology therapy

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2017-08-02 (Actual); Primary Completion 2024-01-05 (Actual); Study Completion 2024-01-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (12):
- China (12):
  - Local Institution - 0015, Beijing, Beijing Municipality
  - Local Institution - 0001, Beijing, Beijing Municipality
  - Local Institution, Guangzhou, Guangdong
  - Local Institution - 0012, Guangzhou, Guangdong
  - Local Institution - 0011, Harbin, Heilongjiang
  - Local Institution, Zhengzhou, Henan
  - Local Institution - 0021, Wuhan, Hubei
  - Local Institution - 0020, Xi'an, Shan1xi
  - Local Institution - 0016, Shanghai, Shanghai Municipality
  - Local Institution - 0018, Chengdu, Sichuan
  - Local Institution - 0004, Tianjin, Tianjin Municipality
  - Local Institution - 0013, Hangzhou, Zhejiang

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Part 1: Arm A: NIVO 3 mg/kg Q2 + IPI 1 mg/kg Q6
- Part 1: Arm B: NIVO 3 mg/kg Q3 + IPI 1 mg/kg Q3
- Part 1: Arm C: NIVO 1 mg/kg Q3 + IPI 3 mg/kg Q3
- Part 2: Arm D: NIVO 3 mg/kg Q3 + IPI 1mg/kg Q3
Period: Overall Study
Arm/Group | Part 1: Arm A | Part 1: Arm B | Part 1: Arm C | Part 2: Arm D
Started | 9 | 9 | 9 | 9
Completed (= completed treatment) | 1 | 4 | 1 | 7
Not Completed | 8 | 5 | 8 | 2
Not completed — Disease Progression | 5 | 4 | 6 | 1
Not completed — Study Drug Toxicity | 2 | 0 | 0 | 1
Not completed — Participant requested to discontinue study treatment | 0 | 1 | 0 | 0
Not completed — Participant Withdrew Consent | 1 | 0 | 0 | 0
Not completed — Maximum Clinical benefit | 0 | 0 | 1 | 0
Not completed — Other Reasons | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: Arm A | Part 1: Arm B | Part 1: Arm C | Part 2: Arm D | Total
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 8 | 8 | 6 | 29
  >=65 years | 2 | 1 | 1 | 3 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4 | 5 | 13
  Male | 8 | 6 | 5 | 4 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 9 | 9 | 9 | 9 | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 9 | 9 | 9 | 9 | 36
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) in Part 1.
Description: Number of participants with Adverse events
Time Frame: From first dose to 100 days post last dose (Approximately on average Arm A: 8.77 Months, Arm B 20.4 Months, Arm C 24.1 Months)
Population: All treated participants in Part 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Arm A | Part 1: Arm B | Part 1: Arm C
Number analyzed (Participants) | 9 | 9 | 9
Participants | 7 | 9 | 9

2. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs) in Part 1.
Description: Number of participants with Adverse events
Time Frame: as for outcome 1
Population: All treated participants in Part 1
Measure: Count of Participants; unit: Participants
Groups:
- Part 1: Arm B: NIVO 3 mg/kg Q3 + IPI 1mg/kg Q3
Arm/Group | Part 1: Arm A | Part 1: Arm B | Part 1: Arm C
Number analyzed (Participants) | 9 | 9 | 9
Participants | 4 | 3 | 3

3. Primary Outcome: Number of Participants With Adverse Events Leading to Discontinuation in Part 1.
Description: Number of participants with Adverse events
Time Frame: as for outcome 1
Population: All treated participants in Part 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Arm A | Part 1: Arm B | Part 1: Arm C
Number analyzed (Participants) | 9 | 9 | 9
Participants | 3 | 0 | 0

4. Primary Outcome: Number of Participants With Adverse Events Leading to Death in Part 1.
Description: Number of participants with Adverse Events leading to death.
Time Frame: as for outcome 1
Population: All treated participants in Part 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Arm A | Part 1: Arm B | Part 1: Arm C
Number analyzed (Participants) | 9 | 9 | 9
Participants | 1 | 1 | 0

5. Primary Outcome: Number of Participants With Clinical Laboratory Abnormalities in Part 1.
Description: Number of participants with clinical laboratory abnormalities.
Time Frame: as for outcome 1
Population: All treated participants in Part 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Arm A | Part 1: Arm B | Part 1: Arm C
Number analyzed (Participants) | 9 | 9 | 9
Participants
  Any Grade | 5 | 9 | 7
  Grade 3-4 | 1 | 4 | 1

6. Primary Outcome: BICR-Assessed ORR in Part 2
Description: ORR is defined as the number of subjects with a best overall response (BOR) of confirmed complete response (CR) or partial response (PR) assessed by BICR, according to RECIST v1.1 criteria, divided by the number of treated subjects.
  The BOR is defined as the best response designation recorded between the date of first dose and the date of initial objectively documented progression per RECIST v1.1 or the date of subsequent therapy, whichever occurs first. For participants without documented progression or subsequent therapy, all available response designations will contribute to the BOR determination. For purposes of analysis, if a subject receives one dose and discontinues the study without assessment or receives subsequent therapy prior to assessment, this participant will be counted in the denominator (as nonrespondent).
Time Frame: between the date of first dose and the date of initial objectively documented progression per RECIST v1.1 or the date of subsequent therapy, whichever occurs first as assessed by BICR. (Approximately on average 3.21 Months)
Population: All treated participants in Part 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part 2: Arm D
Number analyzed (Participants) | 9
Percentage of Participants | 77.8 [40.0 to 97.2]

7. Secondary Outcome: Cmax - Maximum Observed Serum Concentration in Part 1.
Description: Cmax - Maximum observed serum concentration in Part 1.
Time Frame: At Cycle 1 Day 1 and Cycle 3 Day 1 for Arm A, Cycle 1 and Cycle 2 Day 1 for Arm B and C (1 cycle = 42 days)
Population: PK Evaluable Population in Part 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Part 1: Arm A | Part 1: Arm B | Part 1: Arm C
Number analyzed (Participants) | 9 | 9 | 9
ug/mL
  Nivo Cycle 1: number analyzed (Participants) | 9 | 9 | 8
  Nivo Cycle 1 | 59.7 (19) | 69.5 (19) | 22.5 (14)
  Nivo Cycle 2: number analyzed (Participants) | 0 | 8 | 6
  Nivo Cycle 2 |  | 104 (12) | 27.2 (21)
  Nivo Cycle 3: number analyzed (Participants) | 3 | 0 | 0
  Nivo Cycle 3 | 122 (21) |  |
  Ipi Cycle 1: number analyzed (Participants) | 9 | 9 | 8
  Ipi Cycle 1 | 18.9 (18) | 16.8 (43) | 55.0 (33)
  Ipi Cycle 2: number analyzed (Participants) | 0 | 8 | 6
  Ipi Cycle 2 |  | 22.0 (16) | 64.1 (29)
  Ipi Cycle 3: number analyzed (Participants) | 3 | 0 | 0
  Ipi Cycle 3 | 20.1 (17) |  |

8. Secondary Outcome: Tmax - Time of Maximum Observed Serum Concentration in Part 1.
Description: Tmax - Time of maximum observed serum concentration in Part 1.
Time Frame: At Cycle 1 Day 1 and Cycle 3 Day 1 for Arm A, Cycle 1 and Cycle 2 Day 1 for Arm B and C (1 cycle = 42 days)
Population: PK Evaluable Population in Part 1
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1: Arm A | Part 1: Arm B | Part 1: Arm C
Number analyzed (Participants) | 9 | 9 | 9
Hours
  Nivo Cycle 1: number analyzed (Participants) | 9 | 9 | 8
  Nivo Cycle 1 | 1.68 [1.6 to 8.0] | 1.62 [1.5 to 48.0] | 1.59 [1.5 to 1.6]
  Nivo Cycle 2: number analyzed (Participants) | 0 | 8 | 6
  Nivo Cycle 2 |  | 1.55 [1.5 to 47.9] | 4.78 [1.6 to 8.0]
  Nivo Cycle 3: number analyzed (Participants) | 3 | 0 | 0
  Nivo Cycle 3 | 1.65 [1.6 to 8.0] |  |
  Ipi Cycle 1: number analyzed (Participants) | 9 | 9 | 8
  Ipi Cycle 1 | 0.617 [0.5 to 7.0] | 6.83 [0.5 to 46.9] | 0.517 [0.5 to 6.8]
  Ipi Cycle 2: number analyzed (Participants) | 0 | 8 | 6
  Ipi Cycle 2 |  | 6.98 [0.5 to 7.0] | 0.542 [0.5 to 6.9]
  Ipi Cycle 3: number analyzed (Participants) | 3 | 0 | 0
  Ipi Cycle 3 | 6.78 [0.5 to 6.9] |  |

9. Secondary Outcome: AUC(0-T) - Area Under the Plasma Concentration-time Curve in Part 1.
Description: AUC(0-T) - Area under the plasma concentration-time curve from time zero to the last time of the last quantifiable concentration. in Part 1.
Time Frame: At Cycle 1 Day 1 and Cycle 3 Day 1 for Arm A, Cycle 1 and Cycle 2 Day 1 for Arm B and C (1 cycle = 42 days)
Population: PK Evaluable Population in Part 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | Part 1: Arm A | Part 1: Arm B | Part 1: Arm C
Number analyzed (Participants) | 9 | 9 | 9
h*ug/mL
  Nivo Cycle 1: number analyzed (Participants) | 9 | 9 | 8
  Nivo Cycle 1 | 10329 (21) | 14141 (26) | 4056 (25)
  Nivo Cycle 2: number analyzed (Participants) | 0 | 8 | 6
  Nivo Cycle 2 |  | 23348 (28) | 4323 (39)
  Nivo Cycle 3: number analyzed (Participants) | 3 | 0 | 0
  Nivo Cycle 3 | 23147 (31) |  |
  Ipi Cycle 1: number analyzed (Participants) | 9 | 9 | 8
  Ipi Cycle 1 | 2847 (18) | 3377 (27) | 9893 (21)
  Ipi Cycle 2: number analyzed (Participants) | 0 | 8 | 6
  Ipi Cycle 2 |  | 4959 (28) | 11388 (34)
  Ipi Cycle 3: number analyzed (Participants) | 3 | 0 | 0
  Ipi Cycle 3 | 3480 (18) |  |

10. Secondary Outcome: AUC(TAU) - Area Under the Concentration-time Curve in One Dosing Interval in Part 1.
Description: AUC(TAU) - Area under the concentration-time curve in one dosing interval in Part 1.
Time Frame: At Cycle 1 Day 1 and Cycle 3 Day 1 for Arm A, Cycle 1 and Cycle 2 Day 1 for Arm B and C (1 cycle = 42 days)
Population: PK Evaluable Population in Part 1. Inadequate PK Sampling for arm A ipilimumab treatment, so no data was collected
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | Part 1: Arm A | Part 1: Arm B | Part 1: Arm C
Number analyzed (Participants) | 9 | 9 | 9
h*ug/mL
  Nivo Cycle 1: number analyzed (Participants) | 9 | 9 | 8
  Nivo Cycle 1 | 10333 (21) | 13919 (26) | 4002 (19)
  Nivo Cycle 2: number analyzed (Participants) | 0 | 8 | 6
  Nivo Cycle 2 |  | 24467 (23) | 4647 (48)
  Nivo Cycle 3: number analyzed (Participants) | 3 | 0 | 0
  Nivo Cycle 3 | 28098 (18) |  |
  Ipi Cycle 1: number analyzed (Participants) | 0 | 9 | 8
  Ipi Cycle 1 |  | 3339 (27) | 9808 (17)
  Ipi Cycle 2: number analyzed (Participants) | 0 | 8 | 6
  Ipi Cycle 2 |  | 5377 (20) | 12206 (36)
  Ipi Cycle 3: number analyzed (Participants) | 0 | 0 | 0

11. Secondary Outcome: Ceoinf - Serum Concentration Achieved at the End of Study Drug Infusion in Part 1.
Description: Ceoinf - Serum concentration achieved at the end of study drug infusion in Part 1.
Time Frame: At Cycle 1 Day 1 and Cycle 3 Day 1 for Arm A, Cycle 1 and Cycle 2 Day 1 for Arm B and C (1 cycle = 42 days)
Population: PK Evaluable Population in Part 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Part 1: Arm A | Part 1: Arm B | Part 1: Arm C
Number analyzed (Participants) | 9 | 9 | 9
ug/mL
  Nivo Cycle 1: number analyzed (Participants) | 9 | 9 | 8
  Nivo Cycle 1 | 59.4 (19) | 68.4 (21) | 22.5 (14)
  Nivo Cycle 2: number analyzed (Participants) | 0 | 8 | 6
  Nivo Cycle 2 |  | 99.5 (15) | 25.4 (24)
  Nivo Cycle 3: number analyzed (Participants) | 3 | 0 | 0
  Nivo Cycle 3 | 120 (21) |  |
  Ipi Cycle 1: number analyzed (Participants) | 8 | 9 | 8
  Ipi Cycle 1 | 17.7 (26) | 14.0 (50) | 54.8 (33)
  Ipi Cycle 2: number analyzed (Participants) | 0 | 8 | 6
  Ipi Cycle 2 |  | 16.3 (39) | 62.7 (27)
  Ipi Cycle 3: number analyzed (Participants) | 3 | 0 | 0
  Ipi Cycle 3 | 17.1 (33) |  |

12. Secondary Outcome: Ctau - Concentration at the End of Dosing Interval in Part 1.
Description: Ctau - Concentration at the end of dosing interval in Part 1. The Ctau is equivilant to the CTrough at these time points.
Time Frame: At Cycle 1 Day 1 and Cycle 3 Day 1 for Arm A, Cycle 1 and Cycle 2 Day 1 for Arm B and C (1 cycle = 42 days)
Population: PK Evaluable Population in Part 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Part 1: Arm A | Part 1: Arm B | Part 1: Arm C
Number analyzed (Participants) | 9 | 9 | 9
ug/mL
  Nivo Cycle 1: number analyzed (Participants) | 9 | 9 | 8
  Nivo Cycle 1 | 19.7 (24) | 16.0 (32) | 3.46 (32)
  Nivo Cycle 2: number analyzed (Participants) | 0 | 6 | 4
  Nivo Cycle 2 |  | 40.6 (30) | 3.32 (70)
  Nivo Cycle 3: number analyzed (Participants) | 2 | 0 | 0
  Nivo Cycle 3 | 63.2 (24) |  |
  Ipi Cycle 1: number analyzed (Participants) | 9 | 9 | 8
  Ipi Cycle 1 | 4.85 (25) | 3.22 (34) | 8.72 (33)
  Ipi Cycle 2: number analyzed (Participants) | 0 | 5 | 4
  Ipi Cycle 2 |  | 6.74 (24) | 15.4 (27)
  Ipi Cycle 3: number analyzed (Participants) | 3 | 0 | 0
  Ipi Cycle 3 | 6.07 (20) |  |

13. Secondary Outcome: CLT - Total Body Clearance in Part 1.
Description: CLT - Total body clearance in Part 1.
Time Frame: At Cycle 3 Day 1 for Arm A, Cycle 2 Day 1 for Arm B and C (1 cycle = 42 days)
Population: PK Evaluable Population in Part 1 with CLT data collected, Inadequate PK Sampling for arm A nivo/ipilimumab treatment, so no data was collected
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/h
Arm/Group | Part 1: Arm A | Part 1: Arm B | Part 1: Arm C
Number analyzed (Participants) | 3 | 9 | 9
mL/h
  Nivo Cycle 2: number analyzed (Participants) | 0 | 8 | 6
  Nivo Cycle 2 |  | 8.56 (37) | 13.1 (51)
  Nivo Cycle 3: number analyzed (Participants) | 3 | 0 | 0
  Nivo Cycle 3 | 6.99 (16) |  |
  Ipi Cycle 2: number analyzed (Participants) | 0 | 8 | 6
  Ipi Cycle 2 |  | 13.0 (36) | 15.0 (55)
  Ipi Cycle 3: number analyzed (Participants) | 3 | 0 | 0
  Ipi Cycle 3 | NA (NA) — insufficient number of events to produce quantifiable data |  |

14. Secondary Outcome: Css-avg - Average Concentration Over a Dosing Interval (AUC(TAU)/Tau) in Part 1.
Description: Css-avg - Average concentration over a dosing interval (AUC(TAU)/tau) in Part 1.
Time Frame: At Cycle 1 Day 1 and Cycle 3 Day 1 for Arm A, Cycle 1 and Cycle 2 Day 1 for Arm B and C (1 cycle = 42 days)
Population: PK Evaluable Population in Part 1. Inadequate PK Sampling for arm A ipilimumab treatment, so no data was collected
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Part 1: Arm A | Part 1: Arm B | Part 1: Arm C
Number analyzed (Participants) | 9 | 9 | 9
ug/mL
  Nivo Cycle 1: number analyzed (Participants) | 9 | 9 | 8
  Nivo Cycle 1 | 30.8 (21) | 27.6 (26) | 7.94 (19)
  Nivo Cycle 2: number analyzed (Participants) | 0 | 8 | 6
  Nivo Cycle 2 |  | 48.5 (23) | 9.22 (48)
  Nivo Cycle 3: number analyzed (Participants) | 3 | 0 | 0
  Nivo Cycle 3 | 83.6 (18) |  |
  Ipi Cycle 1: number analyzed (Participants) | 0 | 9 | 8
  Ipi Cycle 1 |  | 6.63 (27) | 19.5 (17)
  Ipi Cycle 2: number analyzed (Participants) | 0 | 8 | 6
  Ipi Cycle 2 |  | 10.7 (20) | 24.2 (36)
  Ipi Cycle 3: number analyzed (Participants) | 0 | 0 | 0

15. Secondary Outcome: AI - Accumulation Index in Part 1.
Description: AI - Accumulation index; ratio of an exposure measure at steady-state to that after the first dose (exposure measure includes AUC (TAU) in Part 1.
  Here SS = Steady State Here FD = First Dose
Time Frame: At Cycle 3 Day 1 for Arm A, Cycle 2 Day 1 for Arm B and C (1 cycle = 42 days)
Population: PK Evaluable Population in Part 1. Inadequate PK Sampling for arm A nivo/ipilimumab treatment, so no data was collected
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio of AUC(Tau) at SS vs FD
Arm/Group | Part 1: Arm A | Part 1: Arm B | Part 1: Arm C
Number analyzed (Participants) | 3 | 9 | 9
ratio of AUC(Tau) at SS vs FD
  Nivo Cycle 2: number analyzed (Participants) | 0 | 8 | 6
  Nivo Cycle 2 |  | 1.65 (22) | 1.13 (30)
  Nivo Cycle 3: number analyzed (Participants) | 3 | 0 | 0
  Nivo Cycle 3 | 2.71 (4) |  |
  Ipi Cycle 2: number analyzed (Participants) | 0 | 8 | 6
  Ipi Cycle 2 |  | 1.50 (20) | 1.26 (22)
  Ipi Cycle 3: number analyzed (Participants) | 3 | 0 | 0
  Ipi Cycle 3 | NA (NA) — insufficient number of events to produce quantifiable data |  |

16. Secondary Outcome: T-HALFeff - Effective Elimination Half-life in Part 1.
Description: T-HALFeff - Effective elimination half-life that explains the degree of accumulation observed for a specific exposure measure (exposure measure includes AUC(TAU), Cmax, or Ctau) in Part 1.
Time Frame: At Cycle 3 Day 1 for Arm A, Cycle 2 Day 1 for Arm B and C (1 cycle = 42 days)
Population: PK Evaluable Population in Part 1. Inadequate PK Sampling for arm A nivo/ipilimumab treatment, so no data was collected
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part 1: Arm A | Part 1: Arm B | Part 1: Arm C
Number analyzed (Participants) | 3 | 9 | 9
Hours
  Nivo Cycle 2: number analyzed (Participants) | 0 | 8 | 4
  Nivo Cycle 2 |  | 385 (36) | 263 (37)
  Nivo Cycle 3: number analyzed (Participants) | 3 | 0 | 0
  Nivo Cycle 3 | 507 (4) |  |
  Ipi Cycle 2: number analyzed (Participants) | 0 | 8 | 5
  Ipi Cycle 2 |  | 325 (38) | 282 (14)
  Ipi Cycle 3: number analyzed (Participants) | 3 | 0 | 0
  Ipi Cycle 3 | NA (NA) — insufficient number of events to produce quantifiable data |  |

17. Secondary Outcome: Number of Participants With Nivolumab Anti Drug Antibodies in Part 1.
Description: Number of participants with nivolumab Anti Drug Antibodies in Part 1.
Time Frame: At baseline and from first dose to last dose (Approximately on average of Arm A 24.54 weeks, Arm B 76 weeks, Arm C 92.5 Weeks)
Population: All Treated Subjects with Baseline and at Least One Post-baseline Evaluable ADA Assessment (Part 1)
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Arm A | Part 1: Arm B | Part 1: Arm C
Number analyzed (Participants) | 9 | 9 | 7
Participants
  Baseline ADA Positive | 0 | 2 | 0
  ADA Positive | 0 | 0 | 3
  Neutralizing Positive | 0 | 0 | 1
  ADA Negative | 9 | 9 | 4

18. Secondary Outcome: Number of Participants With Ipilimumab Anti Drug Antibodies in Part 1.
Description: Number of participants with Ipilimumab Anti Drug Antibodies in Part 1.
Time Frame: as for outcome 17
Population: All Treated Subjects with Baseline and at Least One Post-baseline Evaluable ADA Assessment (Part 1)
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Arm A | Part 1: Arm B | Part 1: Arm C
Number analyzed (Participants) | 9 | 9 | 7
Participants
  Baseline ADA Positive | 1 | 0 | 2
  ADA Positive | 0 | 0 | 0
  Neutralizing Positive | 0 | 0 | 0
  ADA Negative | 9 | 9 | 7

19. Secondary Outcome: Investigator-Assessed ORR in Part 2
Description: ORR is defined as the number of subjects with a best overall response (BOR) of confirmed complete response (CR) or partial response (PR) assessed by Investigator, according to RECIST v1.1 criteria, divided by the number of treated subjects.
  The BOR is defined as the best response designation recorded between the date of first dose and the date of initial objectively documented progression per RECIST v1.1 or the date of subsequent therapy, whichever occurs first. For participants without documented progression or subsequent therapy, all available response designations will contribute to the BOR determination. For purposes of analysis, if a subject receives one dose and discontinues the study without assessment or receives subsequent therapy prior to assessment, this participant will be counted in the denominator (as nonrespondent).
Time Frame: between the date of first dose and the date of initial objectively documented progression per RECIST v1.1 or the date of subsequent therapy, whichever occurs first as assessed by the Investigator. (Approximately on average 2 Months)
Population: All treated participants in Part 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part 2: Arm D
Number analyzed (Participants) | 9
Percentage of Participants | 66.7 [29.9 to 92.5]

20. Secondary Outcome: Investigator-Assessed Disease Control Rate (DCR) in Part 2
Description: The percentage of participants whose BOR is confirmed CR or confirmed PR or stable disease (SD) for at least 12 weeks as per investigator.
Time Frame: between the date of first dose and the date of initial objectively documented progression per RECIST v1.1 as assessed by the Investigator. (Approximately on average 5 Months)
Population: All treated participants in Part 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part 2: Arm D
Number analyzed (Participants) | 9
Percentage of Participants | 88.9 [51.8 to 99.7]

21. Secondary Outcome: BICR-Assessed Disease Control Rate (DCR) in Part 2
Description: The percentage of participants whose BOR is confirmed CR or confirmed PR or stable disease (SD) for at least 12 weeks as per BICR.
Time Frame: Approximately 5.92 Months
Population: All treated participants in Part 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part 2: Arm D
Number analyzed (Participants) | 9
Percentage of Participants | 88.9 [51.8 to 99.7]

22. Secondary Outcome: BICR-Assessed Duration of Response (DOR) in Part 2
Description: The time between the date of first confirmed response to the date of the first documented tumor progression (per RECIST 1.1), or death due to any cause, whichever occurs first as per BICR.
Time Frame: From first dose to 100 days post last dose (approximately 102 weeks)
Population: All confirmed responders per BICR in Part 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 2: Arm D
Number analyzed (Participants) | 7
Months | NA [15.21 to NA] — Median and ULN were not reached due to insufficient number of events to calculate via KM methodology.

23. Secondary Outcome: Investigator-Assessed Duration of Response (DOR) in Part 2
Description: The time between the date of first confirmed response to the date of the first documented tumor progression (per RECIST 1.1), or death due to any cause, whichever occurs first as per investigator.
Time Frame: From first dose to 100 days post last dose (approximately 102 weeks)
Population: All confirmed responders per investigator in Part 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 2: Arm D
Number analyzed (Participants) | 6
Months | NA [NA to NA] — Median, LLN and ULN were not reached due to insufficient number of events to calculate via KM methodology.

24. Secondary Outcome: BICR-Assessed Progression Free Survival (PFS) in Part 2
Description: as for outcome 22
Time Frame: From first dose to 100 days post last dose (approximately 102 weeks)
Population: All Treated participtants in Part 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 2: Arm D
Number analyzed (Participants) | 9
Months | NA [1.22 to NA] — Insufficient number of events to calculate median and ULN using Kaplan-Meier methodology.

25. Secondary Outcome: Investigator-Assessed Progression Free Survival (PFS) in Part 2
Description: as for outcome 23
Time Frame: From first dose to 100 days post last dose (approximately 102 weeks)
Population: All Treated participtants in Part 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 2: Arm D
Number analyzed (Participants) | 9
Months | NA [1.22 to NA] — Insufficient number of events to calculate median and ULN using Kaplan-Meier methodology.

ADVERSE EVENTS:
Time Frame: All-Cause mortality, Adverse Events and Serious Adverse Events: From first dose to 100 days post last dose (Approximately on average Arm A: 8.77 Months, Arm B 20.4 Months, Arm C 24.1 Months and Arm D: 23.8 Months.
Description: The number at Risk for All-Cause Mortality represents all Randomized Participants. The number at Risk for Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication
Arm/Group | Part 1: Arm A | Part 1: Arm B | Part 1: Arm C | Part 2: Arm D
All-Cause Mortality (participants affected / at risk) | 2/9 | 2/9 | 1/9 | 1/9
Serious Adverse Events (participants affected / at risk) | 4/9 | 3/9 | 3/9 | 4/9
Other Adverse Events (participants affected / at risk) | 7/9 | 9/9 | 9/9 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Arm A (N=9) | Part 1: Arm B (N=9) | Part 1: Arm C (N=9) | Part 2: Arm D (N=9)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Thyroiditis subacute (Endocrine disorders) | 0 | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Liver injury (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Starvation ketoacidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 1
Completed suicide (Psychiatric disorders) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Arm A (N=9) | Part 1: Arm B (N=9) | Part 1: Arm C (N=9) | Part 2: Arm D (N=9)
Anaemia (Blood and lymphatic system disorders) | 4 | 6 | 2 | 3
Leukocytosis (Blood and lymphatic system disorders) | 1 | 1 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 4 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 2 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 2 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Autoimmune thyroiditis (Endocrine disorders) | 0 | 0 | 1 | 0
Goitre (Endocrine disorders) | 0 | 0 | 1 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 1 | 4 | 1
Hypothyroidism (Endocrine disorders) | 1 | 3 | 3 | 5
Thyroiditis subacute (Endocrine disorders) | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 2 | 3 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 2 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 3 | 3
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 1 | 1
Gastritis erosive (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 2 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 3 | 0
Asthenia (General disorders) | 2 | 2 | 3 | 1
Face oedema (General disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 1
Generalised oedema (General disorders) | 0 | 0 | 0 | 1
Malaise (General disorders) | 0 | 1 | 0 | 1
Mass (General disorders) | 0 | 0 | 1 | 0
Nodule (General disorders) | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 1 | 0 | 1 | 0
Pain (General disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 5 | 2 | 6 | 2
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Liver injury (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 2
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0
Helicobacter infection (Infections and infestations) | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 1
Orchitis (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia fungal (Infections and infestations) | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 2
Face injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Neck injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 3 | 4 | 5
Amylase increased (Investigations) | 0 | 0 | 0 | 2
Anti-thyroid antibody increased (Investigations) | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 3 | 4 | 6
Bacterial test positive (Investigations) | 1 | 0 | 0 | 0
Bilirubin conjugated decreased (Investigations) | 0 | 1 | 0 | 0
Bilirubin conjugated increased (Investigations) | 1 | 2 | 3 | 3
Blood albumin decreased (Investigations) | 1 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 2 | 2 | 4
Blood bilirubin unconjugated increased (Investigations) | 0 | 0 | 0 | 1
Blood calcium decreased (Investigations) | 0 | 1 | 0 | 0
Blood chloride decreased (Investigations) | 2 | 0 | 1 | 0
Blood creatine phosphokinase MB increased (Investigations) | 0 | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 3 | 4 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 1
Blood glucose increased (Investigations) | 0 | 1 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 1
Blood pH increased (Investigations) | 1 | 0 | 0 | 0
Blood potassium decreased (Investigations) | 1 | 1 | 0 | 0
Blood sodium decreased (Investigations) | 2 | 1 | 1 | 0
Blood thyroid stimulating hormone increased (Investigations) | 0 | 0 | 1 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 2
Haematocrit decreased (Investigations) | 2 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 2 | 0 | 2 | 0
Lipase increased (Investigations) | 0 | 1 | 0 | 4
Neutrophil count decreased (Investigations) | 0 | 3 | 0 | 3
Neutrophil count increased (Investigations) | 1 | 0 | 0 | 0
Occult blood positive (Investigations) | 0 | 0 | 0 | 1
Oxygen saturation decreased (Investigations) | 1 | 0 | 0 | 0
PCO2 increased (Investigations) | 1 | 0 | 0 | 0
PO2 decreased (Investigations) | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 1 | 1 | 2
Prealbumin decreased (Investigations) | 0 | 0 | 0 | 1
Protein total decreased (Investigations) | 2 | 0 | 0 | 0
Protein urine present (Investigations) | 0 | 2 | 1 | 0
Red blood cell count decreased (Investigations) | 3 | 0 | 1 | 0
Red blood cells urine positive (Investigations) | 0 | 0 | 2 | 0
Thyroid hormones increased (Investigations) | 0 | 0 | 1 | 0
Thyroxine free decreased (Investigations) | 0 | 0 | 0 | 1
Troponin I increased (Investigations) | 0 | 1 | 0 | 0
Urinary occult blood positive (Investigations) | 0 | 0 | 1 | 0
Urine output decreased (Investigations) | 0 | 0 | 2 | 0
Weight decreased (Investigations) | 0 | 0 | 4 | 1
Weight increased (Investigations) | 2 | 2 | 0 | 2
White blood cell count decreased (Investigations) | 0 | 2 | 0 | 2
White blood cell count increased (Investigations) | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 2 | 4 | 2
Hyperalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypochloraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 2 | 1 | 0
Essential tremor (Nervous system disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0
Bipolar I disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 0 | 1
Oliguria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 4 | 1 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 3 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 2 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 3 | 5 | 2
Rash (Skin and subcutaneous tissue disorders) | 2 | 1 | 2 | 2
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Venous thrombosis limb (Vascular disorders) | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
"AUC(TAU) for ipi in Arm A, Cycle 1 and Cycle 3 could not be reported because there were not enough PK samples collected. Samples were only taken up to 336 hours after dosing, but the full TAU is 1008 hours, so it was not possible to calculate AUC(TAU) for these cycles. In Cycle 2, only a single PK sample was collected (at Week 3, prior to nivo dose administration) for both nivo and ipi. Therefore, AUC(TAU) could not be calculated or reported for nivo and ipi in Arm A, Cycle 2."

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-22): https://cdn.clinicaltrials.gov/large-docs/78/NCT03195478/Prot_SAP_000.pdf